CLINICAL TRIAL: NCT06642961
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Phase II Trail Evaluating the Efficacy and Safety of GR1802 Injection in Patients with Moderate to Severe Asthma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1802-003
Record Dates: First submitted 2024-10-14; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- GR1802 300mg Q2W (Experimental): GR1802 is injected subcutaneously (SC) with a loading dose of 600 mg at the first dose, and then 300 mg each time, once every 2 weeks (Q2W) for a total of 12 doses.
  Interventions: Drug: GR1802 injection
- GR1802 150mg Q2W (Experimental): GR1802 is injected subcutaneously (SC) with a loading dose of 300 mg at the first dose, and then 150 mg each time, once every 2 weeks (Q2W) for a total of 12 doses.
  Interventions: Drug: GR1802 injection
- Placebo (Placebo Comparator): Subcutaneous injection (SC), once every 2 weeks (Q2W) for a total of 12 doses
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GR1802 injection — GR1802 will be administered SC.
  Arms: GR1802 150mg Q2W
Drug: GR1802 injection — GR1802 will be administered SC.
  Arms: GR1802 300mg Q2W
Other: Placebo — The placebo will be administered SC.
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled study to evaluate the efficacy and safety of GR1802 injection in comparison to placebo in patients with atopic dermatitis. Patients will receive GR1802 injection or Placebo every 2 Weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤70 years old, male or female.
2. The subject meet the diagnostic criteria of GINA 2021 requiring a diagnosis of asthma for at least 12 months and fulfilled one of the following criteria:

(1) The subject has received medium-to-high dose ICS combined with at least one control drug, such as LABA, LTRA, theophylline, for at least 3 months before baseline visit, and maintained stable treatment regimen and dosage for at least 1 month before baseline visit; (2) The subject have been on a 3rd controlled drug for at least 3 consecutive months and on a stable dose for ≥1 month prior to baseline visit; (3) The subject must have been on maintenance therapy with ≤10mg/day prednisone or equivalent dose of OCS continuously for at least 3 months and have been receiving therapy at a stable dose for ≥1 month prior to the baseline visit.

3. 35%≤ Pre-bronchodilator FEV1 measured ≤ 80% of the normal predicted value at screening and baseline visits.

4. Asthma Control Questionnaire-5 (ACQ-5) score ≥1.5 at screening and baseline visits.

5. A positive bronchodilation test (≥12% increase in the FEV1 post-bronchodilator and an absolute FEV1 increase of ≥200 mL) within 12 months before screening.

6. Subjects must have experienced at least one severe asthma exacerbation event within 12 months before screening, denfined as: systemic use of glucocorticoids for ≥3 days (at least twice the dose of current use); and/or an emergency visit due to asthma symptoms resulting in hospitalisation, and/or asthma requiring additional systemic glucocorticoid intervention therapy.

7. Willingness to follow the requirements of the study protocol and willingness of the patient or his/her legal representative to sign a written informed consent.

Exclusion Criteria:

1. Chronic obstructive pulmonary disease (COPD) or other lung disease that may impair lung function, as judged by the investigator.
2. Have experienced a severe asthma exacerbation event within 1 month before baseline visit.
3. Lung disease other than asthma with clinically significant impact on efficacy or safety evaluation confirmed by clinical or imaging evidence （e.g., chest X-ray, CT, MRI）within 12 months before baseline visit.
4. Evidence of active tuberculosis infection at screening.
5. Current smokers or former smokers who quit smoking less than 6 months.
6. Former smokers with a smoking history of more than 10 pack-years.
7. Subjects who have history of drug or alcohol abuse (alcohol abuse defined as consumption of more than 28 units of alcohol per week :1 unit = 285 ml of beer or 25 ml of spirits ≥40% alcohol by volume or 1 glass of wine) within 2 years before baseline visit.
8. Long-term reversal of daily sleep patterns (e.g., long-term night shift workers).
9. Subjects who need to be treated with non-selective β1-adrenergic receptor blockers for any reason, or who are on selective β1-blockers but have unstable doses in the 1 month prior to the baseline visit.
10. Underwent an IgE antibody within 130 days prior to the baseline visit, or received prior treatment with an IL-4R antibody (e.g., dupilumab); and those who have received other biologics within 5 half-lives (half-life known) or 6 months (half-life unknown).
11. Treatment with herbs and pCms with asthma-alleviating effects within 4 weeks prior to the baseline visit (except topical herbs).
12. Underwent immunoglobulin (IVIG) therapy, allergen-specific immunotherapy (SIT) within 3 months prior to the baseline visit or plan to be treated with the therapy during the trial.
13. Underwent bronchial thermoplasty within 3years before baseline visit or plan to be treated with the therapy during the trial.
14. Comorbidities requiring ICS (e.g. TB) or LABA (e.g. severe heart disease, insulin-dependent diabetes mellitus, uncontrolled hypertension, hyperthyroidism, etc.) resulting in compromised treatment of the comorbidities.
15. Prolonged QTc interval or ventricular tachycardia requiring pharmacological treatment.
16. Pregnant or lactating women.
17. Positive hepatitis B surface antigen (except for HBVDNA test below 500 IU/ml) and hepatitis B core antibody (except for HBVDNA test below 500 IU/ml) at screening; positive HCV antibody, HIV antibody, and TP-Ab (except for those who are RPR or TRUST negative).
18. Those with existing or suspected acute or chronic infections in the 4 weeks prior to the baseline visit and who have received antibacterial, antiviral, antifungal, antiparasitic or antiprotozoal therapy.
19. Received live or attenuated vaccine within 12 weeks before baseline visit or planned to receive live or attenuated vaccine during the study period.
20. History of vital organ transplantation (e.g. heart, lung, kidney, liver) or haematopoietic stem cell/bone marrow transplantation.
21. Patients with active autoimmune diseases, or autoimmune diseases being treated with immunosuppressive drugs (e.g. inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis, psoriasis, Hashimoto's thyroiditis, Graves' disease).
22. History of severe herpes virus infections, e.g., herpes encephalitis, disseminated herpes.
23. Malignancy within 5 yearsbefore baseline visit (except squamous carcinoma in situ, basal cell carcinoma and cervical carcinoma in situ of the skin, which have been completely treated without any sign of recurrence).
24. Poorly controlled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg. Note: Determined by 2 consecutive elevated readings. If the initial blood pressure reading exceeds this limit, the blood pressure may be re-measured after the subject has rested for ≥10 minutes. If the repeated measurement is below the limit, the second value is acceptable).
25. The following laboratory test abnormalities were present at screening:

    Haemoglobin <10.0 g/dL (100.0 g/L) (men) or <9.0 g/dL (90.0 g/L) (women); white blood cell count <3.0×109/L; neutrophil count <1.5 x 109 /L; platelet count <100 x 109 /L; alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ) > 1.5 times upper limit of normal (ULN); serum creatinine > 1.0 times ULN; total bilirubin > 1.5 times ULN; alkaline phosphatase > 1.5 times ULN.
26. Females and/or males of childbearing potential and their partners who refuse to: use highly effective (female subjects and their partners)/effective (male subjects and their partners) contraception, have a childbearing, egg donation programme (females), or a sperm donation programme (males), from the time of signing the Informed Consent Form until 6 months after the end of the last dose;
27. Participation in another clinical trial treatment within 12 weeks prior to the baseline visit.
28. The investigator considers that there are any conditionswhich are inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pre-bronchodilator FEV1 (forced expiratory volume in 1 second) at 12 weeks. | 12weeks
  Absolute change from baseline in pre-bronchodilator FEV1 in each dose group at 12 weeks of GR1802 treatment compared with placebo.

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator FEV1 at 24 weeks. | 24weeks
  Absolute change from baseline in pre-bronchodilator FEV1 at e24 weeks.
Percent change from baseline in pre-bronchodilator FEV1 at 12 and 24 weeks. | 12weeks and 24weeks
  Percent change from baseline in pre-bronchodilator FEV1 at 12 and 24 weeks.
Annualized rate of subjects experiencing severe asthma exacerbations. | 24weeks and 32weeks
  Annualized rate of subjects experiencing severe asthma exacerbations during the 24-week randomized treatment and throughout the trial period.
Time to the first onset of the severe asthma exacerbation event. | 32weeks
  Time from baseline to the first onset of the severe asthma exacerbation event.
Annualized rate of subjects experiencing the event of loss of asthma control (LOAC). | 24weeks and 32weeks
  Annualized rate of subjects experiencing the event of loss of asthma control (LOAC) during the 24-week randomized treatment and throughout the trial period.
Time to the onset of the first event of LOAC. | 32weeks
  Time from baseline to the onset of the first event of LOAC.
Change from baseline in other lung function measures. | 24weeks
  Changes from baseline in FEV1 percentage of predicted value (FEV1% Pred) and Peak diurnal and nocturnal expiratory flow (PEF)
Changes from baseline in the Asthma Control Questionnaire-5 (ACQ-5)score and ACQ-7 score at each evaluation time point. | 2、4、8、12、16、20、24、28 、32weeks
  The ACQ-5 is a questionnaire used to evaluate the degree of asthma control. Each question is scored from 0 to 6 (on a 7-point scale) according to its severity. The higher the score, the less satisfactory symptom control is.
Change from baseline in the Asthma Quality of Life Questionnaire (AQLQ) score at 12weeks and 24 weeks. | 12weeks and 24weeks
  The AQLQ is a disease-specific health-related quality of life instrument that taps both physical and emotional impact of disease. Scores range 1-7, with higher scores indicating better quality of life.
Total daily use of asthma reliever | 24weeks
  Total daily use of asthma relief medication
Safety evaluation indicators | 32weeks
  Safety evaluation indicators: Adverse Events, Laboratory Tests, Vital Signs, Electrocardiograms, Physical Examination, etc.
Concentration of GR1802 at each evaluation time point. | Baseline up to week 32
  To evaluate the trough concentration at steady-state of GR1802 for each dose group. Population pharmacokinetic analysis is performed using a nonlinear mixed-effects model.
Anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs). | Baseline up to week 32
  Incidence of anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs) (if applicable).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China